CLINICAL TRIAL: NCT03787849
Title: Investigation of the DNA Methylation Profile in Children Who Presented Emergence Delirium
Brief Title: Epigenetics in PostOperative Pediatric Emergence Delirium
Acronym: EPOPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria José Carvalho Carmona, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EPOPED-USP
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Emergence Delirium; Postoperative Complications; DNA Methylation
Keywords: Emergence delirium; Child; Postoperative complications; DNA methylation; Epigenetic
MeSH Terms: conditions — Emergence Delirium; Postoperative Complications | interventions — Sevoflurane; Anesthesia, Inhalation; Propofol; Anesthesia, Intravenous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not aware of anesthesia technique. Outcome assessor of DNA methylation are not aware of anesthesia technique since they will analyze blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Active Comparator): All children will receive inhalation anesthesia with sevoflurane through facial mask in concentrations between 3-8% for anesthesia induction . After induction and peripheral vein puncture, the anesthesia will be maintained only with sevoflurane 3% until completion of the procedure.
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): All children will receive inhalation anesthesia with sevoflurane through facial mask in concentrations between 3-8% until lost of conscience and peripheral vein puncture. After that, sevoflurane will be turned off and its clearance will be analyzed through gas analyzer monitor. From here, anesthesia will be maintained as total venous with continuous propofol infusion 100 mcg.kg.min-1 until completion of the procedure.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — All children will receive inhalation anesthesia with sevoflurane through facial mask in concentrations between 3-8% for anesthesia induction. After induction and peripheral vein puncture, the anesthesia will be maintained only with sevoflurane 3% until completion of the procedure.
  Other Names: Inhalation Anesthesia
  Arms: Sevoflurane
Drug: Propofol — All children will receive inhalation anesthesia with sevoflurane through facial mask in concentrations between 3-8% until lost of conscience and peripheral vein puncture. After that, sevoflurane will be turned off and its clearance will be analyzed through gas analyzer monitor. From here, anesthesia will be maintained as total venous with continuous propofol infusion 100 mcg.kg.min-1 until completion of the procedure.
  Other Names: Intravenous Anesthesia
  Arms: Propofol

SUMMARY:
Emergence delirium (ED) infers the occurrence of behavior and cognition changes during the early postoperative period. Main signs and symptoms of ED are the disturbances of consciousness and awareness of the environment, with disorientation and perceptual alterations, including hypersensitivity to external stimuli and hyperactive motor behaviors. The incidence may be higher than 80%. Risk factors include pre-school age, use of sevoflurane, ophthalmologic and otorhinolaryngologic surgeries, child anxiety, parental or caregiver anxiety. The recurrence of ED is controversial. The only validated scale for diagnosis of ED is the PAED (Pediatric Anesthesia Emergence Delirium). Prevention is the best approach, as well as the use of alpha-2 agonists, propofol and total intravenous anesthesia. There are still no clear markers for postoperative delirium, especially ED. Cognitive alterations may be related to epigenetic modifications. Anesthesia-induced epigenetic changes may be the key to understanding perioperative complications and outcomes and is a field of future research in anesthesia. The study aims to analyze the DNA methylation profile in children with ED. A prospective, randomized study will be carried out in up to 322 children undergoing general anesthesia (inhalation group or intravenous group) to perform endoscopic procedures at the Instituto da Criança, Hospital das Clinicas, Faculdade de Medicina, Universidade de Sao Paulo, Brazil. Patients will have blood samples drawn, and analysis of the DNA methylation profile through the array technique will be performed in 40 children (20 of each group ) who presented ED as well as in 08 control cases. Also, the occurrence of ED will be correlated with the degree of anxiety of the child, parents and during anesthetic induction, in addition to comparing the two anesthetic techniques with the occurrence of ED and late postoperative cognitive alterations.

DETAILED DESCRIPTION:
BACKGROUND: The risks of neurotoxicity and late cognitive impairment supported the recent US Food and Drug Administration (FDA) recommendation on caution in the indication of anesthesia in children up to 3 years of age. Among the cognitive alterations related to pediatric anesthesia, emergence delirium (ED) is frequent in pre-school children. There is no consensus on the risk factors and forms of ED prevention, which occurs more frequently after inhalation anesthesia. On the other hand, anesthesia-induced epigenetic changes may be the key to understanding various complications and perioperative outcomes. There are no specific biomarkers for ED. Such biomarkers would be used to measure the risk of ED and would contribute to prevention and treatment. It has been hypothesized that behavioral changes in ED may be related to epigenetic modifications, analyzed through the DNA methylation profile. OBJECTIVES: The primary aim of the study is to investigate the DNA methylation profile in children with ED. The secondary objectives are to evaluate the correlation between the DNA methylation profile with the anesthetic technique and the degree of preoperative anxiety. METHODS: Children (N=322) from 1 to 12 years old, candidates to digestive endoscopy under general anesthesia will be recruited in an outpatient clinic from a tertiary university hospital. After informed consent, the child and parents' preoperative anxiety will be assessed through the modified Yale Preoperative Anxiety Scale (mYPAS) and VAS-Anx (Anxiety Visual Analogic Scale), respectively. The quality of anesthetic induction will be evaluated through Pediatric Anesthesia Behavior (PAB) scale and Perioperative Adult Child Behavior Interaction Scale (PACBIS). After inhaled induction with sevoflurane, blood sample collection will be performed to evaluate DNA methylation, followed by randomization in two groups to maintain anesthesia using the venous technique, with propofol or inhaled anesthesia with sevoflurane. Upon awakening, the ED will be evaluated through PAED (Pediatric Anesthesia Emergence Delirium) scale. Twenty children from each group presenting ED as well as 08 control cases will have their venous blood samples sent for DNA methylation analysis using the array technique. After hospital discharge, the postoperative behavioral changes will be observed through the PHBQ (Post Hospitalization Behavior Questionnaire) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* children with ASA physical status 1, 2 or 3

Exclusion Criteria:

* children under psychiatric medication
* developmental delays
* genetics syndromes that course with developmental delays
* contraindication to randomization

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
DNA methylation profile of children who presented emergence delirium | An average of one month after discharge from outpatient clinic.
  DNA methylation profile will be measured through an array experiment in the Illumina iScanSQ (Illumina®) platform using the BeadChip Infinium MethylationEPIC and BeadChip HumanCytoSNP850K kits, following the protocol and manufacturer's instructions. The extracted samples will be initially treated with bisulfite using the EZ DNA Methylation Kit (Zymo Research®). The methylation profile is measured by the Beta value. This value ranges from 0 to 1. Closer to zero, more hypomethylated is the DNA and closer to 1, more hypermethylated is the DNA. To compare the profile, the average Beta value of each patient with emergence delirium and their controls will be used. All raw data obtained will be analyzed by bioinformatics methods to compose the DNA methylation profile of each patient.

SECONDARY OUTCOMES:
Emergence delirium | First, 5th, 10th and 15th minutes after anesthesia awakening
  Emergence delirium will be measured through Pediatric Anesthesia Emergence Delirium (PAED) scale. This scale measures 5 items regarding child's awakening: eye contact with the caregiver, purposefulness of child's action, awareness of child's surroundings, child's restlessness and if the child is inconsolable. The first three items are scored from 4 to 1 as follow: 4 not at all, 3 just a little, 2 quite a bit, 1 very much, 0 extremely. Items 4 and 5 are scored as follow: 0 not at all, 1 just a little, 2 quite a bit, 3 very much, 4 extremely. The scores of each item were summed to obtain a total Pediatric Anesthesia Emergence Delirium (PAED) scale score. The degree of emergence delirium increased directly with the total score. We considered a score of ≥ 10 as a cutoff of emergence delirium.
Children's preoperative anxiety | 10 minutes before induction of anesthesia
  This outcome will be measured through modified Yale Preoperative Anxiety Scale (mYPAS). This scale analysis 5 items regarding child's behavior right before induction of anesthesia. A. Activity 1 Looking around. 2 Not exploring. 3 Moving from toy to parent in unfocused manner. 4 Actively trying to get away. B. Vocalizations 1 Reading or asking questions. 2 Responding to adults but whispers. 3 Quiet or no sounds. 4 Whimpering or silently crying. 5 Crying. 6 Crying or screaming loudly. C. Emotional expressivity 1 Manifestly happy. 2 Neutral. 3 Worried to frightened. 4 Distressed. D. State of apparent arousal 1 Alert. 2 Child sitting still and quiet. 3 Vigilant. 4 Panicked. E. Use of parents 1 Busy playing. 2 Reaches out to parent. 3 Looks to parents quietly. 4 Keeps parent. To calculate the final score, we divide each item rating by the highest possible, add all of the produced values, divide by 5, and multiply by 100. Score of ≥ 30 indicates high anxiety before anesthesia.
Caregiver's anxiety before anesthesia | 10 minutes before induction of anesthesia
  This outcome will be measured through a Visual Analogic Scale (VAS) validated for anxiety. This is a 100-mm scale, which will be applied to caregivers right before induction of anesthesia. Score higher than or equal to 70 mm will be considered as high caregiver's anxiety.
Children's behavior and adult interaction during anesthesia induction | First minute during monitoring and anesthesia induction
  This outcome will be measured through Perioperative Adult Child Behavior Interaction Scale (PACBIS). The PACBIS consists of four domains (Child Coping, Child Distress, Parent Positive, and Parent Negative), each of which is assigned one of three possible scores (0, 1 or 2). Scores for each domain are assigned based upon the observer's impression of the most typical expression of the subject's behavior within that domain during the observation period. By identifying the specific area leading to maladaptive behavioral responses, we will be able to correlate with occurrence of emergence delirium.
Children's behavior during anesthesia induction | First minute during anesthesia induction
  This outcome will be measured through Pediatric Anesthesia Behavior (PAB) score. The Pediatric Anesthesia Behavior (PAB) score is scored from one to three based upon the criteria: Group 1 happy calm and controlled, compliant with induction, Group 2 (sad) tearful and/or withdrawn but compliant with induction or Group 3 (mad) loud vocal resistance (screaming or shouting) and/or physical resistance to induction requiring physical restraint by staff and/or parents. Higher scores (2 or 3) could be associated with emergence delirium, and the development of posthospitalization behavior changes.
Post hospitalization behavior changes | First, 7th and 14th day after discharge from outpatient clinic
  This outcome will be measured through Post Hospital Behavior Questionnaire. This questionnaire is composed by the following questions: Does your child make a fuss about eating? Does your child spend time just sitting or lying? Is your child uninterested in what goes on around him/her? Does your child get upset when you leave him/her alone for a few minutes? Does your child need a lot of help doing things? Is it difficult to get your child interested in doing things? Does your child have temper tantrums? Is it difficult to get your child to talk to you? Does your child have bad dreams or wake up and cry? Does your child have trouble getting to sleep? Does your child have a poor appetite? For each item, parents are asked to compare their child's behavior before hospitalization to their current behavior as follows: much less than before (1), less than before (2), same as before (3), more than before (4), and much more than before (5). Score ≥ 3 will be considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Maria JC Carmona, PhD, Principal Investigator — Associate Professor
Locations (1):
- Instituto da Criança do Hospital das Clinicas da FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen TG. Use of anesthetics in young children Consensus statement of the European Society of Anaesthesiology (ESA), the European Society for Paediatric Anaesthesiology (ESPA), the European Association of Cardiothoracic Anaesthesiology (EACTA), and the European Safe Tots Anaesthesia Research Initiative (EuroSTAR). Paediatr Anaesth. 2017 Jun;27(6):558-559. doi: 10.1111/pan.13160. No abstract available. PMID 28474809
- [Background] Andropoulos DB, Greene MF. Anesthesia and Developing Brains - Implications of the FDA Warning. N Engl J Med. 2017 Mar 9;376(10):905-907. doi: 10.1056/NEJMp1700196. Epub 2017 Feb 8. No abstract available. PMID 28177852
- [Background] Mason KP. Paediatric emergence delirium: a comprehensive review and interpretation of the literature. Br J Anaesth. 2017 Mar 1;118(3):335-343. doi: 10.1093/bja/aew477. PMID 28203739
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Locatelli BG, Ingelmo PM, Emre S, Meroni V, Minardi C, Frawley G, Benigni A, Di Marco S, Spotti A, Busi I, Sonzogni V. Emergence delirium in children: a comparison of sevoflurane and desflurane anesthesia using the Paediatric Anesthesia Emergence Delirium scale. Paediatr Anaesth. 2013 Apr;23(4):301-8. doi: 10.1111/pan.12038. Epub 2012 Oct 9. PMID 23043512
- [Background] Jacob Z, Li H, Makaryus R, Zhang S, Reinsel R, Lee H, Feng T, Rothman DL, Benveniste H. Metabolomic profiling of children's brains undergoing general anesthesia with sevoflurane and propofol. Anesthesiology. 2012 Nov;117(5):1062-71. doi: 10.1097/ALN.0b013e31826be417. PMID 22929729
- [Background] Fournier A, Krause R, Winterer G, Schneider R. Biomarkers of postoperative delirium and cognitive dysfunction. Front Aging Neurosci. 2015 Jun 9;7:112. doi: 10.3389/fnagi.2015.00112. eCollection 2015. PMID 26106326
- [Background] Huett C, Baehner T, Erdfelder F, Hoehne C, Bode C, Hoeft A, Ellerkmann RK. Prevention and Therapy of Pediatric Emergence Delirium: A National Survey. Paediatr Drugs. 2017 Apr;19(2):147-153. doi: 10.1007/s40272-017-0212-x. PMID 28130755
- [Background] Somaini M, Engelhardt T, Fumagalli R, Ingelmo PM. Emergence delirium or pain after anaesthesia--how to distinguish between the two in young children: a retrospective analysis of observational studies. Br J Anaesth. 2016 Mar;116(3):377-83. doi: 10.1093/bja/aev552. PMID 26865130
- [Background] Moore AD, Anghelescu DL. Emergence Delirium in Pediatric Anesthesia. Paediatr Drugs. 2017 Feb;19(1):11-20. doi: 10.1007/s40272-016-0201-5. PMID 27798810
- [Background] Almenrader N, Passariello M, Coccetti B, Haiberger R, Pietropaoli P. Premedication in children: a comparison of oral midazolam and oral clonidine. Paediatr Anaesth. 2007 Dec;17(12):1143-9. doi: 10.1111/j.1460-9592.2007.02332.x. PMID 17986032
- [Background] Prabhu MK, Mehandale SG. Comparison of oral dexmedetomidine versus oral midazolam as premedication to prevent emergence agitation after sevoflurane anaesthesia in paediatric patients. Indian J Anaesth. 2017 Feb;61(2):131-136. doi: 10.4103/0019-5049.199852. PMID 28250481
- [Background] El Batawi HY. Effect of preoperative oral midazolam sedation on separation anxiety and emergence delirium among children undergoing dental treatment under general anesthesia. J Int Soc Prev Community Dent. 2015 Mar-Apr;5(2):88-94. doi: 10.4103/2231-0762.155728. PMID 25992332
- [Background] Costi D, Cyna AM, Ahmed S, Stephens K, Strickland P, Ellwood J, Larsson JN, Chooi C, Burgoyne LL, Middleton P. Effects of sevoflurane versus other general anaesthesia on emergence agitation in children. Cochrane Database Syst Rev. 2014 Sep 12;2014(9):CD007084. doi: 10.1002/14651858.CD007084.pub2. PMID 25212274
- [Background] Chandler JR, Myers D, Mehta D, Whyte E, Groberman MK, Montgomery CJ, Ansermino JM. Emergence delirium in children: a randomized trial to compare total intravenous anesthesia with propofol and remifentanil to inhalational sevoflurane anesthesia. Paediatr Anaesth. 2013 Apr;23(4):309-15. doi: 10.1111/pan.12090. PMID 23464658
- [Background] Abdulatif M, Ahmed A, Mukhtar A, Badawy S. The effect of magnesium sulphate infusion on the incidence and severity of emergence agitation in children undergoing adenotonsillectomy using sevoflurane anaesthesia. Anaesthesia. 2013 Oct;68(10):1045-52. doi: 10.1111/anae.12380. Epub 2013 Aug 3. PMID 23909742
- [Background] Levenson JM, Sweatt JD. Epigenetic mechanisms in memory formation. Nat Rev Neurosci. 2005 Feb;6(2):108-18. doi: 10.1038/nrn1604. PMID 15654323
- [Background] Day JJ, Sweatt JD. Epigenetic mechanisms in cognition. Neuron. 2011 Jun 9;70(5):813-29. doi: 10.1016/j.neuron.2011.05.019. PMID 21658577
- [Background] Stary CM, Patel HH, Roth DM. Epigenetics: The Epicenter for Future Anesthesia Research? Anesthesiology. 2015 Oct;123(4):743-4. doi: 10.1097/ALN.0000000000000808. No abstract available. PMID 26259141
- [Background] Block RI, Magnotta VA, Bayman EO, Choi JY, Thomas JJ, Kimble KK. Are Anesthesia and Surgery during Infancy Associated with Decreased White Matter Integrity and Volume during Childhood? Anesthesiology. 2017 Nov;127(5):788-799. doi: 10.1097/ALN.0000000000001808. PMID 28837436
- [Background] Jevtovic-Todorovic V. Exposure of Developing Brain to General Anesthesia: What Is the Animal Evidence? Anesthesiology. 2018 Apr;128(4):832-839. doi: 10.1097/ALN.0000000000002047. PMID 29271804
- [Background] Graham MR. Clinical update regarding general anesthesia-associated neurotoxicity in infants and children. Curr Opin Anaesthesiol. 2017 Dec;30(6):682-687. doi: 10.1097/ACO.0000000000000520. PMID 28915132
- [Background] Warner DO, Shi Y, Flick RP. Anesthesia and Neurodevelopment in Children: Perhaps the End of the Beginning. Anesthesiology. 2018 Apr;128(4):700-703. doi: 10.1097/ALN.0000000000002121. No abstract available. PMID 29533967